CLINICAL TRIAL: NCT06417749
Title: MIND Diet and Cognitive Function in Middle-aged and Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Changzheng Yuan, Research Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LL20240353
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Function; Dementia
Keywords: Cognitive Function; Dietary Pattern
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel design, with one arm being the control arm and the other being the intervention arm (MIND diet education and food supply).
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind design, where the outcome assessors will be masked from the assignment of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Placebo Comparator): General dietary advice
  Interventions: Behavioral: Control arm
- Intervention arm (Active Comparator): MIND diet education
  Interventions: Behavioral: Intervention arm

INTERVENTIONS:
Behavioral: Control arm — Participants will receive a copy of the Chinese Dietary Guidelines leaflet at baseline.
  Arms: Control arm
Behavioral: Intervention arm — Participants will be given three MIND diet education videos on different topics at baseline and during follow-up. In addition, each participant will receive a MIND diet education brochure at baseline and some food supply during follow-up.
  Arms: Intervention arm

SUMMARY:
A 12-month cluster-randomized controlled trial designed to test the effect of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet education on the rate of cognitive change and several other secondary outcomes in 1200 adults aged 40-69 years.

DETAILED DESCRIPTION:
Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet and Cognitive Decline in Middle-aged and Elderly People is a 12-month cluster-randomized controlled trial designed to test the effect of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet education on the rate of cognitive change and several other secondary outcomes in 1200 adults aged 40-69 years. The proposed MIND diet for this study is a hybrid of the Mediterranean and DASH diets but with selected modifications based on the most compelling evidence in the diet-dementia field and Chinese Dietary Guidelines 2022. Specifically, the proposed MIND diet education will emphasize the consumption of whole grains, dark green leafy vegetables, dark red/yellow vegetables, other vegetables, berries and citrus, poultry, fish and seafood, beans and legumes, nuts, olive and seed oils, and green tea, and restrict red and processed meats, animal fat, fried foods, and sweets and pastries. The trial will employ a cluster randomization design comparing the effects on cognitive change of the MIND intervention diet education among 1200 adults aged 40-69 years. Secondary outcomes will include dietary behavior changes, health status changes, etc. The proposed study is sited at Taian, Shandong, China.

ELIGIBILITY:
Inclusion Criteria:

* Normal chewing function, able to eat hard foods such as nuts.
* Willing to participate and sign an informed consent form.
* Able to understand research procedures and adhere to them throughout the entire study period.

Exclusion Criteria:

* Participation in or have participated in other clinical trial studies within the past year.
* Medication to treat Alzheimer's or Parkinson's disease.
* Diagnosis of severe chronic diseases, such as cancer.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in 5-min Montreal Cognitive Assessment (MoCA) score | 12 months
  Cognitive function will be assessed using the MoCA at baseline and during follow-up.

SECONDARY OUTCOMES:
Change in EuroQol Five Dimensions (EQ-5D) scale | 12 months
  The 5-level EQ-5D (EQ-5D-5L) will be used to assess life quality. Evaluations will be conducted at baseline and during follow-up.
Change in 8-Item Alzheimer's Diseases Screening Tool (AD-8) score | 12 months
  AD-8 will be used to assess cognitive function. Evaluations will be conducted at baseline and during follow-up.
Change in Mediterranean-Dietary Approach to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) diet score | 12 months
  Dietary behavior will be assessed using food frequency questionnaire (FFQ). A 15-point MIND diet score will be calculated to reflect the MIND diet adherence among both groups of participants. Evaluations will be conducted at baseline and during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Mutiple Counties, Taian, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Interested collaborators may put in a request.